CLINICAL TRIAL: NCT02467777
Title: Comparison of Forced Air and Conductive Patient Heating Systems During Ambulatory Surgeries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fox Valley Orthopedic Institute (Other)
Responsible Party: Principal Investigator, Vishal Mehta, Orthopaedic Surgeon, Fox Valley Orthopedic Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15-025
Record Dates: First submitted 2015-04-23; First posted 2015-06-10 (Estimated); Results first posted 2017-03-23 (Actual); Last update posted 2017-05-11 (Actual); Status verified 2017-04

CONDITIONS: Hypothermia
Keywords: orthopaedics; post-operative warming
MeSH Terms: conditions — Hypothermia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Forced Air (Active Comparator): Bair Hugger
  Interventions: Device: Bair Hugger
- Conductive Warming (Active Comparator): VitaHeat
  Interventions: Device: VitaHeat

INTERVENTIONS:
Device: Bair Hugger
  Arms: Forced Air
Device: VitaHeat
  Arms: Conductive Warming

SUMMARY:
Comparison of forced air and conductive warming devices in outpatient orthopaedic surgeries.

DETAILED DESCRIPTION:
Patients will be randomized into either the Forced Air group (FA) or Conductive Heat group (CH). Randomization will be based on computer-generated codes that will be maintained in sequentially numbered opaque envelopes. Fifty patients will be recruited with 25 patients being randomized into each group.

In patients assigned to the FA group, a Bair Hugger (Arizant Medical, Inc., Eden Prairie, Minnesota) forced-air cover will be positioned over the upper body (if lower extremity surgery) or lower body (if upper extremity surgery). The forced-air blower will be set and activated per standard practice usually after prepping and draping.

In patients assigned to the CH group, a VitaHeat (VitaHeat, Inc, Aurora, IL) conductive heating device will be placed under the torso of the patient. The device will be set and activated per standard practice usually just after positioning of the patient on the operating table.

Patients in both groups will be otherwise draped per surgical routine. Ambient temperature will be maintained near 20°C. Temperatures will be recorded using a temporal artery thermometer.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing orthopaedic outpatient surgeries over 18 years old

Exclusion Criteria:

* allergic to material of bair hugger

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-06; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Fox Valley Orthopedics, Geneva, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Forced Air | Conductive Warming
Started | 23 | 27
Completed | 23 | 27
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Forced Air | Conductive Warming | Total
Number analyzed (Participants) | 23 | 27 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 19 | 20 | 39
  >=65 years | 4 | 7 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 53 (11.52) | 50.4 (16.15) | 51.6 (14.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 11 | 18
  Male | 16 | 16 | 32
Region of Enrollment [Number; unit: participants]
  United States | 23 | 27 | 50

OUTCOME MEASURES:

1. Primary Outcome: Temperature
Description: Measured by temporal artery thermometer
Time Frame: Intra-Operative
Measure: Mean (Standard Deviation); unit: degrees celsius
Arm/Group | Forced Air | Conductive Warming
Number analyzed (Participants) | 23 | 27
degrees celsius | 97.95 (.60) | 97.64 (.58)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Forced Air | Conductive Warming
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/27
Other Adverse Events (participants affected / at risk) | 0/23 | 0/27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No